CLINICAL TRIAL: NCT02339987
Title: Procure Tumor and Initiate Melanoma Tumor-Reactive Tumor Infiltration
Status: Terminated | Type: Observational
Why Stopped: original PI left institute, no plan to continue using samples
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TIL-PROCURE-0614
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue from resection of a metastatic melanoma lesion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Procure Tumor and Initiate Melanoma Tumor-Reactive Tumor Infiltration Lymphocytes (TIL)

DETAILED DESCRIPTION:
The purpose of this study is to allow the collection of tissue from subjects to be used in future research studies by scientists and to isolate tumor fighting cells for the future treatment of Melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have metastatic melanoma with a resectable metastasis who are undergoing resection for palliation, therapeutic or curative purpose.
2. Patients must be > 15 years of age and must have metastatic melanoma.
3. Patients must meet standard pre-operative requirements as determined by the surgeon to be candidates for surgery.
4. Patients must be able to understand and sign the Informed Consent document.
5. Patients must be able to complete the supplemental data form

Exclusion Criteria:

1. women who are pregnant or breastfeeding
2. inability to give consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cancer clinic
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Evaluate Feasibility of conducting TIL procurement in a single-site setting | 5 years
  Cell viability, viable number and TIL potency using standardized methods
Evaluate Safety of conducting TIL procurement in a single-site setting | 5 separate TIL procedures
  lab personnel training during procurement, isolation, testing tumor reactivity and cryopreservation

SECONDARY OUTCOMES:
To determine whether TIL Procurement, isolation, testing tumor reactivity and cryopreservation can be performed at John Wayne Cancer Institute (JWCI) and Providence Saint John's Health Center (PSJHC) and infused into patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No